CLINICAL TRIAL: NCT00405496
Title: Phase 2a Study of 0.05% Difluprednate Ophthalmic Emulsion in the Treatment of Anterior Uveitis (Inluding Iritis, Cyclitis, Iridocyclitis, and Panuveitis).
Brief Title: Study of Difluprednate Ophthalmic Emulsion in the Treatment of Uveitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sirion Therapeutics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SJE2079/2-02-PC
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Last update posted 2006-11-30 (Estimated); Status verified 2006-11

CONDITIONS: Anterior Uveitis
MeSH Terms: conditions — Uveitis, Anterior

INTERVENTIONS:
Drug: Difluprednate Ophthalmic Emulsion

SUMMARY:
The purpose of this phase 2 study is to determine if difluprednate ophthalmic emulsion is effective in the treatment of uveitis.

DETAILED DESCRIPTION:
The primary objective was to investigate the efficacy and safety of 0.05% difluprednate ophthalmic emulsion in patients with endogenous anterior uveitis and to determine its clinical usefulness for treatment of this disease in the early phase of development, in comparison with Rinderon® solution (containing 0.1% betamethasone sodium phosphate) that has widely been used for treatment of postoperative inflammation, uveitis, etc. as a steroid ophthalmic solution.

The secondary objective was to establish the evaluation system for a dose-finding study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with endogenous anterior uveitis (including panuveitis)
* Patients with 20 or more anterior chamber cell within one field of the aqueous humor (Grade 3 or higher in clinical signs and grading) as measured with a slitlamp microscope
* Patients aged ≥20 years and <75 years who could clearly express their subjective symptoms (Patients aged 20 years at giving informed consent were included in the study.)
* Patients giving written informed consent prior to initiation of the study

Exclusion Criteria:

* Patients who did not meet all of the above inclusion criteria
* Patients receiving systemic administration or topical administration to the head or face including instillation of corticosteroid, nonsteroidal anti-inflammatory drugs, antiphlogistic enzymes, immunosuppressive drugs or colchicines within 1 week before the initial instillation of the study drug
* Patients with glaucoma or ocular hypertension (IOP ≥21 mmHg)
* Patients with corneal erosion or corneal ulcer
* Patients with viral keratoconjunctival diseases, tuberculos eye diseases, fungal eye diseases or bacterial eye diseases
* Patients with diabetes mellitus
* Patients with allergy to corticosteroids
* Patients requiring use of contact lens during the study period
* Women who were or might be pregnant
* Patients participating in other clinical studies within 6 months before initiation of the present study
* Patients with sensitivity to steroids(Patients who previously exhibited increased IOP after instillation of a steroid ophthalmic solution)
* Patients with fibrins to such an extent that might affect measurement of flare

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2000-03; Study Completion 2001-04

PRIMARY OUTCOMES:
The anterior chamber cell score was compared between baseline and after completion of the
study treatment (14 +/- 2 days). The efficacy was evaluated with a 4-point scale based on the
reduction of anterior chamber cell.

SECONDARY OUTCOMES:
The overall efficacy was evaluated with a 4-point-scale based on the change in the flare value
(baseline/after completion of the study treatment ratio), as measured with a laser flare cell
meter, and those in anterior chamber flare as measured with a slitlamp microscope and clinical
signs and symptoms after completion of the study treatment (142 days) from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Kanjiro Masudo, Study Chair — Director, Kanto Rosai Hospital